CLINICAL TRIAL: NCT02459314
Title: Comparison of the Efficacy of Plant Sterol-Enriched Soymilk Versus Plain Soymilk in Volunteers With High LDL-Cholesterol
Acronym: sterols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Supawan Buranapin, Assistant Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dutchmill 002
Record Dates: First submitted 2015-05-15; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- soymilk (Placebo Comparator): Soymilk (SM) contained 5 gm soy protein and 6.5 gm sugar per 180 mL package.
  Interventions: Dietary Supplement: soymilk
- sterol/fiber-enriched soymilk (Active Comparator): PLant sterol and soluble fiber-enriched soymilk (SFSM) contained 1 gm free plant sterol, 5 gm inulin (soluble fiber), 5 gm soy protein and 6.5 gm sugar per 180 mL package
  Interventions: Dietary Supplement: plant sterol and soluble fiber-enriched soymilk

INTERVENTIONS:
Dietary Supplement: plant sterol and soluble fiber-enriched soymilk — Sterols compete with LDL-C for absorption in GI tract. A meta-analysis of 41 trials indicated that an intake of 2 g sterols/stanols reduces the LDL-C level by 10%. Additive effects occur when sterols are combined with statins; the combination being more efficacious than a 2 times up-dosing of statins alone. Soluble dietary fibers also have significant cholesterol lowering effects. In a meta-analysis, Brown et al estimate that a daily soluble fiber intake ranging from 9-30 g/d, were associated with 10.6% reduction in LDL-C levels.
  Arms: sterol/fiber-enriched soymilk
Dietary Supplement: soymilk — Soy protein is another LDL-C and total cholesterol lowering food. A meta-analysis by Reynolds K et al. discovered that volunteers receiving 20 to more than 61 g of soy protein had reductions in total cholesterol by 5.26 mg/dL (95% CI -7.14 to -3.38), and LDL-C by 4.25 mg/dL (95% CI -6.00 to -2.50), with an increase of HDL-C by 0.77 mg/dL (95% CI 0.20 to 1.34). Reductions in LDL cholesterol were larger in hypercholesterolemic than in normocholesterolemic subjects.
  Arms: soymilk

SUMMARY:
This was a multicenter, prospective, randomized, double-blinded, controlled-trial study in hypercholesterolemic volunteers (serum LDL-C > 130 mg/dL). Eligible subjects were randomized to receive either plant sterol and soluble fiber-enriched soymilk or plain soymilk 360 mL/day (2 packages a day) for 8 weeks. Venous blood samples were collected from the eligible subjects during pre-treatment (screening period; day -7), every 2 week after treatment (at the end of week 2, 4, 6 and 8) to test for lipid profiles and fasting blood sugar (FBS).

DETAILED DESCRIPTION:
This was a multicenter, prospective, randomized, double-blinded, controlled-trial study in hypercholesterolemic volunteers (serum LDL-C > 130 mg/dL). After initial assessment at the screening period, eligible subjects were randomized to receive either plant sterol and soluble fiber-enriched soymilk (SFSM) or plain soymilk (SM) 360 mL/day (2 packages a day) for 8 weeks. The participants might take the study product as snack, the first one in the morning and the second one in the afternoon. It was possible to take it before or after meal, however taken before meal was highly suggested. A physical examination (including vital signs, height, weight, body mass index, waist circumference, and systemic evaluation) was performed at each visit, every 2 weeks. Concurrent medications usage were record at each visit during the study as well.

Three-day per week of food intake and weekly exercises were recorded and evaluated at every visit. It was recommended every participant to follow dietary control and lifestyle modification to improve hypercholesterolemia during the entire study. Details of overall product satisfaction were evaluated by the participants after 2 and 8 weeks of study products consumption (at visit 2 and 5). To evaluate compliance, the participants were asked to collect and return the empty packages to the investigator every 2 weeks at visit 2, 3, 4, and 5. More than 90% of study product consumption would be considered as eligible on-going subjects.

Venous blood samples were collected from the eligible subjects during pre-treatment (screening period; day -7), every 2 week after treatment (visit 2, 3, 4, 5; at the end of week 2, 4, 6 and 8) to test for lipid profiles and fasting blood sugar (FBS). Adverse events, if any, were recorded immediately after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age > 18 years
2. If female, subject is either post-menopausal or surgically sterilized, or has a negative urine pregnancy test within 7 days prior to enrollment and will use adequate contraception during the study
3. Has LDL-C > 130 mg/dL
4. If subject has been treated with cholesterol-lowering agents prior to admission, he/she must have taken medication regularly at a stable dose for at least 8 weeks
5. Provided written informed consent prior to admission to the study.

Exclusion criteria:

1. Has history of organ transplantation
2. Hypersensitivity to soy bean or has specific allergy to the ingredients of soymilk
3. Has taken any medication that affects serum cholesterol level, such as oral contraceptive pills, high dose diuretics or beta-blockers, antiretroviral protease inhibitors, tegretol, and anabolic steroids, unless these drugs have been consumed at the same dosage for > 8 weeks prior to admission of the study
4. Has serum triglyceride ≥ 400 mg/dL
5. Immunocompromised status, including a debilitated state or malignancy
6. Has consumed any immunosuppressive agents such as cyclosporine, tacrolimus, azathioprine, and chemotherapeutic agents
7. Active liver, renal or thyroid diseases
8. Recent myocardial infarction or stroke within 3 months prior to admission
9. Has recently been admitted in the hospital due to any illness within 2 months prior to admission
10. Frequent alcoholic consumption > 2 a week; with beer > 360 mL, alcohol > 45 mL, wine > 150 mL for female, or beer > 720 mL, whisky > 90 mL, wine > 300 mL for male each time
11. HasGI symptoms such as nausea, vomiting, loss of appetite, premature satiety, diarrhea, or chronic constipation
12. Consume study product less than 90% during in treatment period
13. Pregnancy or breast feeding woman
14. Has previously been admitted to this study
15. Lack of ability or willingness to give informed consent
16. Start taking any medication that may affect serum lipid profiles or immunosuppressive agents during in the study
17. Receiving dietary supplement with plant sterols/ stanols and/ or fiber.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
the change of serum LDL-C levels between 8-week ingestion of plant sterol and soluble fiber-enriched soymilk (SFSM) versus plain soymilk (SM). | 8 weeks
  compare the change of LDL-C between those who took SFSM and those who took SM and between baseline and after 8 weeks of consumption

SECONDARY OUTCOMES:
changes in other lipid profiles (total cholesterol, HDL-C and triglyceride) | 8 weeks
  to evaluate the change of total cholesterol, triglyceride, HDL-C, FBS between SFSM and SM group and between baseline and after 8 weeks of consumption
scale of study product satisfaction | 8 weeks
  score the product satisfaction after 2 weeks and 8 weeks consumption
evaluate any adverse events | 8 weeks
  gastrointestinal side effects of the product consumption

OTHER OUTCOMES:
fasting plasma glucose (FPG) | 8 weeks
  compare the FPG between SFSM and soymilk consumption in 8 weeks and compare between baseline and after 8 weeks of consumption

CONTACTS AND LOCATIONS:
Overall Officials: Supawan Buranapin, MD, Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Clinical trial Unit, Faculty of Medicine, Chiang Mai University, Muang, ChiangMai, Thailand